CLINICAL TRIAL: NCT07283627
Title: Exploring the Evolution of Quality of Life and Emotional Distress Among Cancer Patients Participating in Mind-body Therapies
Acronym: MBT & cancer
Status: Enrolling by invitation | Type: Observational
Sponsor: La Tour Hospital (Other)
Collaborators: OTIUM foundation (Unknown)
Responsible Party: Principal Investigator, Anthony Pernoud, Clinical Project Manager, La Tour Hospital
Other Study IDs: 2025-00543
Record Dates: First submitted 2025-12-04; First posted 2025-12-16 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Cancer; Mind-Body Therapies
Keywords: Cancer; Supportive care; Patient-reported outcomes; Emotional distress; Mind-body therapies; Quality of life; Mindfulness; Laughter yoga; Art therapy; Integrative oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OTIUM Minb-body therapy cohort: This cohort includes adult cancer patients participating in one specific mind-body therapy (MBT) offered at the OTIUM Centers in Geneva and Meyrin. Eligible participants take part in a structured program-mindfulness, laughter yoga, or art therapy-delivered in a group format over approximately 8 to 10 weeks. The cohort is designed to evaluate changes in quality of life and emotional distress associated with participation in the selected MBT. All participants complete standardized patient-reported outcome measures (EORTC QLQ-C30 and HADS) before and after the therapy.

SUMMARY:
Cancer incidence is increasing worldwide, and although survival rates have improved thanks to advances in treatment and early detection, many patients continue to experience reduced quality of life (QoL), anxiety, depression, and distress. Mind-body therapies (MBTs)-including mindfulness, laughter yoga, and art therapy-are increasingly integrated into supportive oncology care. Evidence suggests these therapies may improve psychosocial well-being; however, existing research often suffers from methodological limitations, small samples, and limited generalizability.

The OTIUM centers in Geneva and Meyrin offer structured MBT programs to cancer patients. This project aims to evaluate the evolution of QoL and emotional distress in patients participating in one of these therapies, using validated patient-reported outcome measures (PROMs).

DETAILED DESCRIPTION:
Cancer is one of the leading causes of disease burden, morbidity, and mortality worldwide. With both the aging and growth of the population, combined with overall socioeconomic development, the prominence of cancer is increasing, with an estimated annual incidence of 35 million cases projected by 2050. Advancements in early detection and treatments have improved survival rates and life expectancy, allowing individuals to live with cancer for longer periods of time. However, this life-threatening disease and its treatments may lead to a reduced quality of life (QoL), heightened anxiety, distress and depression. Patients with diagnosed cancer are 28% more likely to experience any mental disorder within a 12-month period compared to the general population (odds ratio: 1.28, 95% confidence interval (CI), 1.14-1.45). The somatic symptoms of cancer such as fatigue, pain, and loss of appetite along with the associated mental health burden, have consistently been associated with higher mortality rates.

Improved cancer survival rates have shifted attention toward the patient's symptom burden, encompassing both physical and mental aspects. Over the past two decades, this has led to the emergence of a holistic care approach. Integrative oncology, defined by the Society of Integrative Oncology, comprises mind and body therapies (MBTs), natural products, and/or lifestyle modifications. MBTs are defined as practices that "focus on the interactions among the brain, mind, body, and behavior, with the intent to use the mind to affect physical functioning and promote health", and have recently been recommended by the Society of Integrative Oncology and American Society of Clinical Oncology guidelines. Such practices comprise, among other, techniques like mindfulness, yoga, art therapy, relaxation or taichi. In this project, the investigators aim to specifically investigate three MBTs: (i) Mindfulness, (ii) Laughter Yoga, and (iii) Art therapy.

* Mindfulness is defined as non-judgmental attention to experiences of the present moment, including thoughts, emotions, and bodily sensations.
* Laughter yoga combines unconditional laughter with yoga breathing practices and yoga stretching poses so that patients laugh different from jokes or humor programs.
* Art therapy is defined as "a form of psychotherapy that uses art media as its primary mode of communication".

To better understand the benefits of therapy for patients, standardized patient-reported outcome measures (PROMs) are increasingly utilized in cancer research. These tools offer valuable insights from the patient's perspective, capturing information on quality of life (QoL) as well as the status of physical, mental, and social health domains. Among the most widely used PROMs in cancer research are the Core Quality of Life Questionnaire developed by the European Organisation for Research and Treatment of Cancer (EORTC QLQ-C30) and the Hospital Anxiety and Depression Scale (HADS), although many other tools are also available. Mindfulness, Laughter Yoga and Art therapy have each proven effective in alleviating depression, anxiety, pain and other symptoms. Adoption of these practices, however, remains limited, likely due to the lack of robustness and diversity of the studies. Indeed, most studies involved a small sample size, with methodological differences in the intervention, with the bulk of the research focusing on women with breast cancer.

Therefore, the purpose of our pragmatic research is to explore and describe the evolution of quality of life and emotional distress in cancer patients participating in one of three mind-body therapies (MBTs), as measured by the EORTC QLQ-C30 and HADS.

According to Art.7 HRO this research project falls under Risk Category A, as the only procedure deviating from routine practice is the collection of standardized PROMs.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with cancer
* Acceptance and signature of an informed consent form
* Age of majority
* Completion of one of the therapies concerned.

Exclusion Criteria:

* Withdrawal of the signed informed consent form
* Metastatic cancer
* Cancer recurrence
* Drugs use against stress
* Memory disorders
* History or current use of a MBT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be selected from individuals receiving supportive oncology services at the OTIUM Centers located in Geneva and Meyrin, Switzerland. These centers provide mind-body therapies as part of routine integrative care for adults living with or recovering from cancer. Patients typically come from the greater Geneva region and may be referred by oncologists at Hôpital de La Tour or may self-present to the centers to participate in non-pharmacological supportive programs. The study population therefore reflects a real-world clinical population engaged in mind-body therapies within an outpatient supportive care setting.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life | From enrollment to the end of treatment at (approximately) 8 weeks
  The primary variable of interest is the total score on the EORTC QLQ-C30, measured at baseline and at the end of treatment, on average 8 weeks after start of treatment. The EORTC QLQ-C30 is scored on a 0 to 100 scale, with higher scores indicating better quality of life for the global health status/quality of life scale. This outcome was selected because it is the most widely used PROM, which facilitates interpretation and comparison with existing literature, and enables us to better assess the quality of care we provide.

SECONDARY OUTCOMES:
Emotional distress | From enrollment to the end of treatment at (approximately) 8 weeks
  The secondary variable of interest is the HADS total score, also measured at the start and end of treatment. The HADS total score ranges from 0 to 42, with higher scores indicating greater psychological distress. Similarly, this outcome was chosen as it is widely used in cancer research and its accuracy has been proven.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Pernoud, MSc, Study Chair — La Tour Hospital
Locations (1):
- La Tour Hospital, Meyrin, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided